CLINICAL TRIAL: NCT04058977
Title: Redefining Survivorship: POWER to Maximize Physical Function for Survivors of Critical Illness: A Randomized Controlled Trial
Brief Title: Redefining Survivorship: POWER to Maximize Physical Function for Survivors of Critical Illness
Acronym: POWER
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawn prior to participant enrollment due to funding status
Sponsor: Kirby Mayer (Other)
Collaborators: Nathan Johnson, PT, PhD (Unknown); Ashley Montgomery-Yates, MD (Unknown); Amy Pastva, PT, PhD (Unknown); Peter E. Morris, MD (Unknown)
Responsible Party: Sponsor-Investigator, Kirby Mayer, Graduate Research Assistant, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 46072
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Critical Illness; Muscle Atrophy or Weakness
MeSH Terms: conditions — Critical Illness; Muscular Atrophy; Asthenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Personnel performing outcomes will be blinded to study group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Power training (Experimental): Randomized to early power training with standardized exercise progression plus standard of care
  Interventions: Other: Power training
- Standard of Care (No Intervention): Standard of care

INTERVENTIONS:
Other: Power training — Progressive exercise protocol with focus on velocity of movement
  Arms: Power training

SUMMARY:
Patients surviving critical illness experience significant skeletal muscle dysfunction and weakness. Muscle atrophy suffered during critical illness has a long-term impact on the functionality and mobility of these individuals. As a result, individuals surviving critical illness have a significant reduction in quality of life, even up to 5 years post discharge. Research including large randomized controls demonstrates that rehabilitation focused on active mobilization may positively influence patient outcomes. Thus, early mobilization is an important intervention that has many purported benefits. Current rehabilitation practice in the intensive care unit (ICU) and recommendations from clinical practice guidelines such as the Society of Critical Care Medicine, PADIS Guidelines support these interventions to reduce the detrimental effects of immobilization during critical illness. Early mobilization is routinely thought of as standard of care for patients admitted for acute respiratory distress syndrome and sepsis. However, a significant number of recent randomized controlled trials implementing early rehabilitation and mobilization interventions fail to demonstrate immediate or long-term benefits.10,11,18,19 Interesting, active mobilization and rehabilitation analyzed in systematic review had no impact on mortality and "no consistent effects of function, quality of life and ICU or hospital length of stay."18 There are a few potential explanations for interventions not leading to reduction in impairment or functional benefit.

Scientific Premise: From our preliminary data (Figure 1) and my clinical experience, a significant cause of the physical impairments in these patients is reductions in muscular power. Muscular power is a critical determinant of functional mobility.20 Preliminary data demonstrate that lower extremity muscle power is significantly reduced in this population and furthermore, these deficits are strongly correlated to physical function. Muscle power training is a potential therapeutic intervention that could lead to more robust improvements in physical function. This concept has been explored extensively in community-dwelling older adults. A recent systematic review of controlled trials demonstrates that power training is superior to traditional resistance training at improving functional performance when comparing the two training modalities.21 Furthermore, power training is feasible for older adults and clinical populations of Parkinson's Disease, Stroke, and frailty.22-27 Thus the feasibility and pragmatic nature of power training is not a concern. Of interest, a randomized controlled trial was completed in institutionalized frail nonagenarians (>85 years or older).27 In this study, no patients drop-out of study due to power training and significant benefits in function were achieved.27 Therefore, the investigators propose a interventional trial to study the effect of a standardized muscle power training program for patients admitted to the ICU for critical illness.

ELIGIBILITY:
Inclusion Criteria:

* admitted to medicine ICU
* acute respiratory failure or ARDS
* sepsis
* anticipated >48 hours MV

Exclusion Criteria:

* acute neurologic infarct
* non-ambulatory prior to hospitalization
* pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Short Performance Physical Battery | 6-month follow-up
  This outcome measure is scored from 0-12 with lower scores representing disability and higher scores representing better physical function. This test has three components including balance, chair rise time, and habitual gait speed. There is a pre-defined scoring system with participants scoring 0-4 on each test, higher representing better function.
  These individual components can then be further analysed based on continuous variables of five repetitions of chair rise and habitual 4-meter gait speed. Faster times to complete the the chair-rise test and faster gait speed represents better physical function.

SECONDARY OUTCOMES:
Quality of life: Eq-5D | 6-month follow-up
  The Eq-5d is a validate quality of life questionnaire that the participant completes. It has five components each on a scale from 1 to 5, which higher scores representing poor or worse quality of life. A total score can be assessed out of possible 25.
Six minute walk test (6-mwt) | 6-month follow-up
  The 6-mwt is a test of physical function and strength in which participant walks as far as possible in six-minutes. Final distance is analysed as a continuous variable with higher distances being better.

CONTACTS AND LOCATIONS:
Overall Officials: Kirby P Mayer, DPT, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Following completion of the proposed experiments, data sharing will be accomplished in a timely fashion via dissemination through publications in peer-reviewed journals and through presentations at national and international meetings.